CLINICAL TRIAL: NCT00289900
Title: A Multicenter, Randomized, Double-Blind, Parallel Group, 12 Week Study to Evaluate the Efficacy and Safety of MK0524B Versus Atorvastatin in Patients With Mixed Hyperlipidemia
Brief Title: Lipid Efficacy and Safety in Participants With Mixed Hyperlipidemia (MK-0524B-024)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0524B-024; MK-0524B-024 (Other: Merck Study Number); 2005_103
Record Dates: First submitted 2006-02-07; First posted 2006-02-10 (Estimated); Results first posted 2016-01-26 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Mixed Hyperlipidemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Atorvastatin; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- MK-0524B 2g/20 mg (Experimental): Co-administration of one tablet of MK-0524A (Extended Release [ER] niacin/laropiprant [LRPT] 1g + one tablet of simvastatin 10 mg for 4 weeks, then co-administration of two tablets of MK-0524A 1g + simvastatin 20 mg for 8 weeks
  Interventions: Drug: MK-0524A; Drug: Simvastatin
- MK-0524B 2g/40mg (Experimental): Co-administration of one tablet of MK-0524A 1g + one tablet of simvastatin 20 mg for 4 weeks, then co-administration of two tablets of MK-0524A 1g + simvastatin 40 mg for 8 weeks
  Interventions: Drug: MK-0524A; Drug: Simvastatin
- Atorvastatin 10 mg (Active Comparator): Atorvastatin 10 mg, orally, once daily for 12 weeks
  Interventions: Drug: Atorvastatin
- Atorvastatin 20 mg (Active Comparator): Atorvastatin 20 mg, orally, once daily for 12 weeks
  Interventions: Drug: Atorvastatin
- Atorvastatin 40 mg (Active Comparator): Atorvastatin 40 mg, orally, once daily for 12 weeks
  Interventions: Drug: Atorvastatin
- Atorvastatin 80 mg (Active Comparator): Atorvastatin 80 mg, orally, once daily for 12 weeks
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: MK-0524A
  Arms: MK-0524B 2g/20 mg; MK-0524B 2g/40mg
Drug: Atorvastatin
  Other Names: Lipitor
  Arms: Atorvastatin 10 mg; Atorvastatin 20 mg; Atorvastatin 40 mg; Atorvastatin 80 mg
Drug: Simvastatin
  Other Names: Zocor
  Arms: MK-0524B 2g/20 mg; MK-0524B 2g/40mg

SUMMARY:
This is a 12-week clinical trial in participants with mixed hyperlipidemia to study the effects of MK-0524B on lipids.The primary hypothesis is that MK-0524B (dosed as MK-0524A coadministered with simvastatin) will be superior to atorvastatin on decreasing the low denisity lipoprotein cholesterol (LDL-C)/high-density lipoprotein cholesterol (HDL-C) ratio for the following dose comparisons: 2g/20 mg MK-0524B versus 10 mg atorvastatin, 2g/40 mg MK-0524B versus 20 mg atorvastatin, 2g/40 mg MK-0524B versus 40 mg atorvastatin, and 2g/40 mg MK-0524B versus 80 mg atorvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Participant 18 to 80 years of age with Mixed Hyperlipidemia with LDL-C between 130 and 190 mg/dL and Triglycerides between 150 and 500 mg/dL

Exclusion Criteria:

* Pregnant or lactating women, or women intending to become pregnant
* Diabetes mellitus that is poorly controlled, newly diagnosed, or taking new or recently adjusted antidiabetic therapy (with the exception of ± 10 units of insulin)
* Human immunodeficiency virus (HIV) positive
* Any of the following within the past 3 months: heart attack, stoke, heart bypass surgery, unstable angina, angioplasty
* Active or chronic liver disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2340 (Actual)
Dates: Start 2006-01-24 (Actual); Primary Completion 2010-08-06 (Actual); Study Completion 2010-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Chen F, Maccubbin D, Yan L, Sirah W, Chen E, Sisk CM, Davidson M, Blomqvist P, McKenney JM. Lipid-altering efficacy and safety profile of co-administered extended release niacin/laropiprant and simvastatin versus atorvastatin in patients with mixed hyperlipidemia. Int J Cardiol. 2013 Jul 15;167(1):225-31. doi: 10.1016/j.ijcard.2011.12.103. Epub 2012 Feb 4. PMID 22305632
- Available data/document: CSR Synopsis Link — http://www.merck.com/clinical-trials/study.html?id=0524B-024&kw=0524B-024&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MK-0524B 2g/20 mg | MK-0524B 2g/40mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Atorvastatin 40 mg | Atorvastatin 80 mg
Started | 297 | 436 | 298 | 439 | 437 | 433
Treated | 297 | 435 | 298 | 439 | 437 | 433
Completed | 229 | 316 | 265 | 380 | 392 | 372
Not Completed | 68 | 120 | 33 | 59 | 45 | 61
Not completed — Adverse Event | 28 | 40 | 13 | 19 | 20 | 33
Not completed — Lost to Follow-up | 7 | 7 | 8 | 8 | 4 | 8
Not completed — Participant had flushing | 18 | 42 | 1 | 2 | 0 | 4
Not completed — Other | 0 | 0 | 0 | 5 | 1 | 0
Not completed — Participant moved | 1 | 0 | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 10 | 21 | 8 | 18 | 12 | 11
Not completed — Protocol Violation | 3 | 9 | 2 | 6 | 7 | 4
Not completed — site terminated | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Not treated | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-0524B 2g/20 mg | MK-0524B 2g/40mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Atorvastatin 40 mg | Atorvastatin 80 mg | Total
Number analyzed (Participants) | 297 | 436 | 298 | 439 | 437 | 433 | 2340
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (10.8) | 55.0 (10.3) | 53.7 (10.6) | 54.8 (10.8) | 55.1 (10.1) | 54.7 (10.5) | 54.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 237 | 169 | 248 | 232 | 258 | 1309
  Male | 132 | 199 | 129 | 191 | 205 | 175 | 1031

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in the LDL-C/HDL-C Ratio
Description: Blood samples taken at baseline and after 12 weeks of treatment to determine the LDL-C and HDL-C levels. The LDL-C/HDL-C ratio was then calculated for baseline and Week 12 and the change from baseline at Week 12 was recorded.
Time Frame: Baseline and Week 12
Population: All randomized participants who had taken at least 1 dose of post-randomization study medication and had a baseline value and at least one post-titration measurement for the endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | MK-0524B 2g/20 mg | MK-0524B 2g/40mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Atorvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 255 | 361 | 280 | 402 | 410 | 402
Percentage Change | -50.9 [-53.8 to -47.9] | -53.0 [-55.4 to -50.7] | -37.6 [-40.5 to -34.8] | -42.4 [-44.5 to -40.0] | -47.9 [-50.1 to -45.7] | -48.8 [-51.1 to -46.6]
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg vs Atorvastatin 10 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Model with factors for baseline LDL-C and triglyceride stratum, gender, cohort of participants, treatment group and baseline parameter covariate; Difference in Least Squares Mean = -13.2, 95% CI 2-sided [-16.8 to -9.6]
Statistical Analysis 2: Comparison: MK-0524B 2g/40mg vs Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = -10.8, 95% CI 2-sided [-13.8 to -7.8]
Statistical Analysis 3: Comparison: MK-0524B 2g/40mg vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = -5.1, 95% CI 2-sided [-8.1 to -2.1]
Statistical Analysis 4: Comparison: MK-0524B 2g/40mg vs Atorvastatin 80 mg; Test type: Superiority or Other; p = 0.007, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = -4.2, 95% CI 2-sided [-7.2 to -1.2]

2. Secondary Outcome: Percentage Change From Baseline in HDL-C
Description: Blood samples taken at baseline and after 12 weeks of treatment to determine the HDL-C levels. The change from baseline at Week 12 was recorded.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | MK-0524B 2g/20 mg | MK-0524B 2g/40mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Atorvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 255 | 361 | 280 | 402 | 410 | 402
Percentage change | 26.9 [24.7 to 29.1] | 26.6 [24.8 to 28.4] | 7.0 [4.8 to 9.1] | 5.3 [3.6 to 7.0] | 4.5 [2.8 to 6.2] | 3.6 [1.9 to 5.3]
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg vs Atorvastatin 10 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = 19.9, 95% CI 2-sided [17.2 to 22.6]
Statistical Analysis 2: Comparison: MK-0524B 2g/40mg vs Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = 21.3, 95% CI 2-sided [19.0 to 23.6]
Statistical Analysis 3: Comparison: MK-0524B 2g/40mg vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = 22.1, 95% CI 2-sided [19.8 to 24.4]
Statistical Analysis 4: Comparison: MK-0524B 2g/40mg vs Atorvastatin 80 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = 23.0, 95% CI 2-sided [20.7 to 25.3]

3. Secondary Outcome: Percentage Change From Baseline in Triglycerides (TG)
Description: Blood samples taken at baseline and after 12 weeks of treatment to determine the TG levels. The change from baseline at Week 12 was recorded.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Percentage change
Arm/Group | MK-0524B 2g/20 mg | MK-0524B 2g/40mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Atorvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 255 | 361 | 280 | 402 | 410 | 402
Percentage change | -40.3 [-44.2 to -36.5] | -42.0 [-45.7 to -38.4] | -21.9 [-25.0 to -18.8] | -23.8 [-26.5 to -21.2] | -30.4 [-32.8 to -27.9] | -33.8 [-36.4 to -31.2]
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg vs Atorvastatin 10 mg; Test type: Superiority or Other; p < 0.001, Non-parametric ANOVA; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -17.3, 95% CI 2-sided [-21.2 to -13.3] — Hodges-Lehmann estimate of the difference between treatments with a corresponding distribution-free confidence interval (CI) based on Wilcoxon's rank sum test
Statistical Analysis 2: Comparison: MK-0524B 2g/40mg vs Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, Non-parametric ANOVA; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -15.5, 95% CI 2-sided [-19.1 to -11.9] — Hodges-Lehmann estimate of the difference between treatments with a corresponding distribution-free CI based on Wilcoxon's rank sum test
Statistical Analysis 3: Comparison: MK-0524B 2g/40mg vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, Non-parametric ANOVA; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -10.3, 95% CI 2-sided [-13.7 to -7.0] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 4: Comparison: Atorvastatin 40 mg vs Atorvastatin 80 mg; Test type: Superiority or Other; p < 0.001, Non-parametric ANOVA; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -6.8, 95% CI 2-sided [-10.2 to -3.4] — [estimate comment as in outcome 3, analysis 2]

4. Secondary Outcome: Percentage Change From Baseline in Non-HDL-C
Description: Blood samples taken at baseline and after 12 weeks of treatment to determine the non-HDL-C levels. The change from baseline at Week 12 was recorded.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | MK-0524B 2g/20 mg | MK-0524B 2g/40mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Atorvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 255 | 361 | 280 | 402 | 410 | 402
Percentage change | -40.4 [-42.9 to -37.9] | -42.2 [-44.2 to -40.2] | -31.3 [-33.7 to -28.9] | -36.8 [-38.7 to -34.9] | -42.6 [-44.5 to -40.7] | -44.6 [-46.6 to -42.7]
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg vs Atorvastatin 10 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = -9.1, 95% CI 2-sided [-12.1 to -6.0]
Statistical Analysis 2: Comparison: MK-0524B 2g/40mg vs Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = -5.4, 95% CI 2-sided [-8.0 to -2.9]
Statistical Analysis 3: Comparison: MK-0524B 2g/40mg vs Atorvastatin 40 mg; Test type: Superiority or Other; p = 0.771, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = 0.4, 95% CI 2-sided [-2.2 to 2.9]
Statistical Analysis 4: Comparison: MK-0524B 2g/40mg vs Atorvastatin 80 mg; Test type: Superiority or Other; p = 0.065, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = 2.4, 95% CI 2-sided [-0.2 to 5.0]

5. Secondary Outcome: Percentage Change From Baseline in LDL-C
Description: Blood samples taken at baseline and after 12 weeks of treatment to determine the LDL-C levels. The change from baseline at Week 12 was recorded.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | MK-0524B 2g/20 mg | MK-0524B 2g/40mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Atorvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 255 | 361 | 280 | 402 | 410 | 402
Percentage change | -40.4 [-43.0 to -37.7] | -42.8 [-44.9 to -40.7] | -33.6 [-36.1 to -31.0] | -39.8 [-41.8 to -37.8] | -45.6 [-47.6 to -43.6] | -47.5 [-49.5 to -45.5]
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg vs Atorvastatin 10 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in least Squares Mean = -6.8, 95% CI 2-sided [-10.2 to -3.5]
Statistical Analysis 2: Comparison: MK-0524B 2g/40mg vs Atorvastatin 20 mg; Test type: Superiority or Other; p = 0.037, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = -3.0, 95% CI 2-sided [-5.8 to -0.2]
Statistical Analysis 3: Comparison: MK-0524B 2g/40mg vs Atorvastatin 40 mg; Test type: Superiority or Other; p = 0.047, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = 2.8, 95% CI 2-sided [0.0 to 5.6]
Statistical Analysis 4: Comparison: MK-0524B 2g/40mg vs Atorvastatin 80 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Sqaures Mean = 4.7, 95% CI 2-sided [2.0 to 7.5]

6. Secondary Outcome: Percentage Change From Baseline in Apolipoprotein (Apo) B
Description: Blood samples taken at baseline and after 12 weeks of treatment to determine the Apo B levels. The change from baseline at Week 12 was recorded.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | MK-0524B 2g/20 mg | MK-0524B 2g/40mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Atorvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 248 | 350 | 272 | 396 | 404 | 389
Percentage change | -36.1 [-38.4 to -33.7] | -38.0 [-39.9 to -36.2] | -26.9 [-29.2 to -24.6] | -32.8 [-34.6 to -31.0] | -37.2 [-38.9 to -35.4] | -38.3 [-40.1 to -36.5]
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg vs Atorvastatin 10 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = -9.2, 95% CI 2-sided [-12.1 to -6.3]
Statistical Analysis 2: Comparison: MK-0524B 2g/40mg vs Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = -5.2, 95% CI 2-sided [-7.7 to -2.8]
Statistical Analysis 3: Comparison: MK-0524B 2g/40mg vs Atorvastatin 40 mg; Test type: Superiority or Other; p = 0.476, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = -0.9, 95% CI 2-sided [-3.3 to 1.5]
Statistical Analysis 4: Comparison: MK-0524B 2g/40mg vs Atorvastatin 80 mg; Test type: Superiority or Other; p = 0.845, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = 0.2, 95% CI 2-sided [-2.2 to 2.7]

7. Secondary Outcome: Percentage Change From Baseline in Apo A-I
Description: Blood samples taken at baseline and after 12 weeks of treatment to determine the Apo A-I levels. The change from baseline at Week 12 was recorded.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | MK-0524B 2g/20 mg | MK-0524B 2g/40mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Atorvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 248 | 350 | 272 | 396 | 404 | 389
Percentage change | 10.7 [8.7 to 12.6] | 8.2 [6.7 to 9.7] | 1.7 [-0.2 to 3.5] | 0.4 [-1.0 to 1.9] | -0.8 [-2.2 to 0.7] | -2.5 [-3.9 to -1.0]
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg vs Atorvastatin 10 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = 9.0, 95% CI 2-sided [6.6 to 11.4]
Statistical Analysis 2: Comparison: MK-0524B 2g/40mg vs Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = 7.7, 95% CI 2-sided [5.8 to 9.7]
Statistical Analysis 3: Comparison: MK-0524B 2g/40mg vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = 9.0, 95% CI 2-sided [7.0 to 10.9]
Statistical Analysis 4: Comparison: MK-0524B 2g/40mg vs Atorvastatin 80 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = 10.7, 95% CI 2-sided [8.7 to 12.7]

8. Secondary Outcome: Percentage Change From Baseline in Total Cholesterol (TC)
Description: Blood samples taken at baseline and after 12 weeks of treatment to determine the TC levels. The change from baseline at Week 12 was recorded.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | MK-0524B 2g/20 mg | MK-0524B 2g/40mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Atorvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 255 | 361 | 280 | 402 | 410 | 402
Percentage change | -28.1 [-30.1 to -26.2] | -30.0 [-31.5 to -28.4] | -24.6 [-26.4 to -22.7] | -29.4 [-30.9 to -27.9] | -34.2 [-35.7 to -32.7] | -36.1 [-37.6 to -34.6]
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg vs Atorvastatin 10 mg; Test type: Superiority or Other; p = 0.003, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = -3.6, 95% CI 2-sided [-6.0 to -1.2]
Statistical Analysis 2: Comparison: MK-0524B 2g/40mg vs Atorvastatin 20 mg; Test type: Superiority or Other; p = 0.595, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = -0.5, 95% CI 2-sided [-2.5 to 1.5]
Statistical Analysis 3: Comparison: MK-0524B 2g/40mg vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = 4.2, 95% CI 2-sided [2.2 to 6.2]
Statistical Analysis 4: Comparison: MK-0524B 2g/40mg vs Atorvastatin 80 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = 6.1, 95% CI 2-sided [4.1 to 8.1]

9. Secondary Outcome: Percentage Change From Baseline in Lipoprotein (a) (Lp[a])
Description: Blood samples taken at baseline and after 12 weeks of treatment to determine the Lp(a) levels. The change from baseline at Week 12 was recorded.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Percentage change
Arm/Group | MK-0524B 2g/20 mg | MK-0524B 2g/40mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Atorvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 248 | 350 | 272 | 396 | 404 | 391
Percentage change | -15.2 [-19.9 to -10.6] | -14.6 [-17.9 to -11.4] | 0.0 [-2.9 to 2.9] | 0.0 [-3.4 to 3.4] | 7.8 [4.6 to 11.1] | 8.8 [5.5 to 12.1]
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg vs Atorvastatin 10 mg; Test type: Superiority or Other; p < 0.001, Non-parametric ANOVA; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -18.8, 95% CI 2-sided [-24.2 to -14.2] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 2: Comparison: MK-0524B 2g/40mg vs Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, Non-parametric ANOVA; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -20.5, 95% CI 2-sided [-25.0 to -16.6] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: MK-0524B 2g/40mg vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, Non-parametric ANOVA; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -23.9, 95% CI 2-sided [-27.8 to -19.4] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 4: Comparison: MK-0524B 2g/40mg vs Atorvastatin 80 mg; Test type: Superiority or Other; p < 0.001, Non-parametric ANOVA; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -24.6, 95% CI 2-sided [-28.6 to -20.0] — [estimate comment as in outcome 3, analysis 2]

10. Secondary Outcome: Percentage Change From Baseline in C-reactive Protein (CRP)
Description: Blood samples taken at baseline and after 12 weeks of treatment to determine the CRP levels. The change from baseline at Week 12 was recorded.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Percentage change
Arm/Group | MK-0524B 2g/20 mg | MK-0524B 2g/40mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Atorvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 246 | 351 | 274 | 397 | 406 | 396
Percentage change | -15.4 [-23.8 to -7.0] | -20.0 [-27.3 to -12.7] | -19.5 [-26.2 to -12.8] | -28.6 [-34.2 to -22.9] | -33.3 [-38.0 to -28.6] | -38.1 [-43.1 to -33.1]
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg vs Atorvastatin 10 mg; Test type: Superiority or Other; p = 0.500, Non-parametric ANOVA; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -0.8, 95% CI 2-sided [-9.6 to 7.5] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 2: Comparison: MK-0524B 2g/40mg vs Atorvastatin 20 mg; Test type: Superiority or Other; p = 0.083, Non-parametric ANOVA; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 6.9, 95% CI 2-sided [0.0 to 13.8] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: MK-0524B 2g/40mg vs Atorvastatin 40 mg; Test type: Superiority or Other; p = 0.005, Non-parametric ANOVA; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 11.9, 95% CI 2-sided [5.2 to 18.8] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 4: Comparison: MK-0524B 2g/40mg vs Atorvastatin 80 mg; Test type: Superiority or Other; p < 0.001, Non-parametric ANOVA; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 16.4, 95% CI 2-sided [9.8 to 22.8] — [estimate comment as in outcome 3, analysis 2]

11. Secondary Outcome: Percentage Change From Baseline in TC/HDL-C Ratio
Description: Blood samples taken at baseline and after 12 weeks of treatment to determine the TC and HDL-C levels. The TC/HDL-C ratio was then calculated for baseline and Week 12 and the change from baseline at Week 12 was recorded.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | MK-0524B 2g/20 mg | MK-0524B 2g/40mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Atorvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 255 | 361 | 280 | 402 | 410 | 402
Percentage change | -41.0 [-43.2 to -38.7] | -42.3 [-44.2 to -40.5] | -28.2 [-30.4 to -26.0] | -31.5 [-33.3 to -29.8] | -36.0 [-37.7 to -34.2] | -36.7 [-38.5 to -35.0]
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg vs Atorvastatin 10 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = -12.8, 95% CI 2-sided [-15.6 to -9.9]
Statistical Analysis 2: Comparison: MK-0524B 2g/40mg vs Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = -10.8, 95% CI 2-sided [-13.2 to -8.4]
Statistical Analysis 3: Comparison: MK-0524B 2g/40mg vs Atorvastatin 40 mg; Test type: Superiority or Other; p = 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = -6.4, 95% CI 2-sided [-8.8 to -4.0]
Statistical Analysis 4: Comparison: MK-0524B 2g/40mg vs Atorvastatin 80 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = -5.6, 95% CI 2-sided [-8.0 to -3.2]

12. Secondary Outcome: Percentage of Participants With Consecutive Elevations in Alanine Aminotransferase (ALT) and/or Aspartate Aminotransferase (AST) of >=3 x Upper Limit of Normal (ULN)
Description: Participants had AST and ALT levels assessed throughout the 12 week treatment period. Participants who had 2 consecutive assessments of either AST or ALT that were 3 x ULN or greater were recorded. The AST UNLs for males and females were 43 U/L and 36 U/L, respectively. The ALT UNLs for males and females were 40 U/L and 33 U/L, respectively.
Time Frame: up to 12 weeks
Population: All participants who had taken at least 1 dose of study medication and had data available for endpoint. Results for participants who received either MK-0524B 2g/20mg or 2g/40 mg were pooled. Results for participants who received atorvastatin 10, 20, 40, or 80 mg were pooled.
Measure: Number; unit: Percentage of Participants
Groups:
- MK-0524B 2g/20 mg and MK-0524B 2g/40mg (Pooled): Participants who received either MK-0524B 2g/20mg or MK-0524B 2g/40mg (pooled)
- Atorvastatin 10, 20, 40, or 80 mg (Pooled): Participants who received either atorvastatin 10, 20, 40 or 80 mg (pooled)
Arm/Group | MK-0524B 2g/20 mg and MK-0524B 2g/40mg (Pooled) | Atorvastatin 10, 20, 40, or 80 mg (Pooled)
Number analyzed (Participants) | 701 | 1577
Percentage of Participants | 0.4 | 1.8
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg and MK-0524B 2g/40mg (Pooled) vs Atorvastatin 10, 20, 40, or 80 mg (Pooled); Test type: Superiority or Other; p = 0.008, Miettinen and Nurminen; Difference in Proportion = -1.4, 95% CI 2-sided [-2.3 to -0.5]

13. Secondary Outcome: Percentage of Participants With Elevations in ALT and/or AST of >=5 x ULN
Description: Participants had AST and ALT levels assessed throughout the 12 week treatment period. Participants who had an assessment of either AST or ALT that was 5 x ULN or greater were recorded. The AST UNLs for males and females were 43 U/L and 36 U/L, respectively. The ALT UNLs for males and females were 40 U/L and 33 U/L, respectively.
Time Frame: up to 12 weeks
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-0524B 2g/20 mg and MK-0524B 2g/40mg (Pooled) | Atorvastatin 10, 20, 40, or 80 mg (Pooled)
Number analyzed (Participants) | 701 | 1577
Percentage of Participants | 0.1 | 0.9
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg and MK-0524B 2g/40mg (Pooled) vs Atorvastatin 10, 20, 40, or 80 mg (Pooled); Test type: Superiority or Other; p = 0.042, Miettinen and Nurminen; Difference in Proportion = -0.7, 95% CI 2-sided [-1.4 to -0.0]

14. Secondary Outcome: Percentage of Participants With Elevations in ALT and/or AST of >=10 x ULN
Description: Participants had AST and ALT levels assessed throughout the 12 week treatment period. Participants who had an assessment of either AST or ALT that was 10 x ULN or greater were recorded. The AST UNLs for males and females were 43 U/L and 36 U/L, respectively. The ALT UNLs for males and females were 40 U/L and 33 U/L, respectively.
Time Frame: up to 12 weeks
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Groups:
- MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled): Participants who received either MK-0524B 2g/20mg or MK-0524B 2g/40mg (pooled)
Arm/Group | MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) | Atorvastatin 10, 20, 40, or 80 mg (Pooled)
Number analyzed (Participants) | 701 | 1577
Percentage of Participants | 0.0 | 0.1
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) vs Atorvastatin 10, 20, 40, or 80 mg (Pooled); Test type: Superiority or Other; p = 0.346, Miettinen and Nurminen; Difference in Proportion = -0.1, 95% CI 2-sided [-0.5 to 0.4]

15. Secondary Outcome: Percentage of Participants With Creatine Kinase (CK) >=10 x ULN
Description: Participants had CK assessed throughout the 12 week treatment period. Participants who had any CK level that was >=10 x ULN were recorded. The UNLs for males and females were 207 U/L and 169 U/L, respectively.
Time Frame: up to 12 weeks
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) | Atorvastatin 10, 20, 40, or 80 mg (Pooled)
Number analyzed (Participants) | 701 | 1577
Percentage of Participants | 0.1 | 0.1
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) vs Atorvastatin 10, 20, 40, or 80 mg (Pooled); Test type: Superiority or Other; p = 0.556, Miettinen and Nurminen; Difference in Proportion = 0.1, 95% CI 2-sided [-0.2 to 0.7]

16. Secondary Outcome: Percentage of Participants With CK >=10 x ULN With Muscle Symptoms
Description: Participants had CK assessed throughout the 24 week treatment period. Participants who had any CK level that was >=10 x ULN and had associated muscle symptoms present within +/- 7 days were recorded. The UNLs for males and females were 207 U/L and 169 U/L, respectively.
Time Frame: up to 12 weeks
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) | Atorvastatin 10, 20, 40, or 80 mg (Pooled)
Number analyzed (Participants) | 701 | 1577
Percentage of Participants | 0.1 | 0.0
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) vs Atorvastatin 10, 20, 40, or 80 mg (Pooled); Test type: Superiority or Other; p = 0.134, Miettinen and Nurminen; Difference in Proportion = 0.1, 95% CI 2-sided [-0.1 to 0.8]

17. Secondary Outcome: Percentage of Participants With CK >=10 x ULN With Muscle Symptoms - Drug Related
Description: Participants had CK assessed throughout the 12 week treatment period. Participants who had any CK level that was >=10 x ULN and had associated muscle symptoms present within +/- 7 days that were reported as at least possibly related to study drug were recorded. The UNLs for males and females were 207 U/L and 169 U/L, respectively.
Time Frame: up to 12 weeks
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) | Atorvastatin 10, 20, 40, or 80 mg (Pooled)
Number analyzed (Participants) | 701 | 1577
Percentage of Participants | 0.1 | 0.0
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) vs Atorvastatin 10, 20, 40, or 80 mg (Pooled); Test type: Superiority or Other; p = 0.134, Miettinen and Nurminen; Difference in Proportion = 0.1, 95% CI [-0.1 to 0.8]

18. Secondary Outcome: Percentage of Participants With New Diagnosis of Impaired Fasting Blood Glucose
Description: Participants had blood glucose levels assessed throughout the 12 week treatment period. Participants who had the new diagnosis of impaired fasting blood glucose were recorded. A pre-defined set of MedDRA terms was used to identify participants whose glycemic status became 'impaired' during the course of treatment (from clinical adverse experience reports). The MedDRA terms were as follows: blood glucose increased, blood glucose abnormal, glucose tolerance decreased, glucose tolerance test abnormal, carbohydrate tolerance decreased, glucose tolerance impaired, hyperglycaemia, impaired fasting glucose, impaired insulin secretion, metabolic syndrome, insulin resistance, insulin resistance syndrome.
Time Frame: up to 12 weeks
Population: All participants who had taken at least 1 dose of study medication and normal glycemic status at baseline. Results for participants who received either MK-0524B 2g/20mg or 2g/40 mg were pooled. Results for participants who received atorvastatin 10, 20, 40, or 80 mg were pooled.
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) | Atorvastatin 10, 20, 40, or 80 mg (Pooled)
Number analyzed (Participants) | 605 | 1343
Percentage of Participants | 0.2 | 0.1
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) vs Atorvastatin 10, 20, 40, or 80 mg (Pooled); Test type: Superiority or Other; p = 0.5625, Miettinen and Nurminen; Difference in Percentage = 0.1, 95% CI 2-sided [-0.3 to 0.9]

19. Secondary Outcome: Percentage of Participants With New Diagnosis of Diabetes
Description: Participants had blood glucose levels assessed throughout the 12 week treatment period. Participants who with newly diagnosed of diabetes were recorded. A participant was classified as having new onset diabetes if they experienced an adverse Event (AE) related to a diagnosis of diabetes (based on a pre-defined set of Medical Dictionary for Regulatory Activities [MedDRA] terms), or if they started taking an anti-diabetic medication during the course of the study. The MedDRA terms were as follows: diabetes mellitus, diabetes mellitus insulin-dependent, diabetes mellitus non-insulin dependent, insulin-requiring type II diabetes mellitus, insulin resistant diabetes, diabetes with hyperosmolarity, latent autoimmune diabetes in adults.
Time Frame: up to 12 weeks
Population: All participants who had taken at least 1 dose of study medication and did not have diabetes at baseline. Results for participants who received either MK-0524B 2g/20mg or 2g/40 mg were pooled. Results for participants who received atorvastatin 10, 20, 40, or 80 mg were pooled.
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) | Atorvastatin 10, 20, 40, or 80 mg (Pooled)
Number analyzed (Participants) | 703 | 1523
Percentage of Participants | 0.9 | 0.2
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) vs Atorvastatin 10, 20, 40, or 80 mg (Pooled); Test type: Superiority or Other; p = 0.0233, Miettinen and Nurminen; Difference in Percentage = 0.7, 95% CI 2-sided [0.1 to 1.7]

20. Secondary Outcome: Percentage of Participants With a Confirmed Adjudicated Cardiovascular Event
Description: Select serious adverse cardiovascular events and all-cause mortality that occurred during the treatment phase of the study were adjudicated by an expert committee external to the sponsor. Those events confirmed by the committee a cardiovascular events were recorded.
Time Frame: up to 14 weeks
Population: All participants who had taken at least 1 dose of study medication. Results for participants who received either MK-0524B 2g/20mg or 2g/40 mg were pooled. Results for participants who received atorvastatin 10, 20, 40, or 80 mg were pooled.
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) | Atorvastatin 10, 20, 40, or 80 mg (Pooled)
Number analyzed (Participants) | 732 | 1607
Percentage of Participants | 0.1 | 0.2
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) vs Atorvastatin 10, 20, 40, or 80 mg (Pooled); Test type: Superiority or Other; p = 0.7858, Miettinen and Nurminen; Difference in Percentage = -0.1, 95% CI 2-sided [-0.4 to 0.6]

21. Secondary Outcome: Percentage of Participants Who Experience at Least 1 Clinical Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. A clinical AE was an AE reported as a result of a clinical examination or reported by the participant.
Time Frame: up to 14 weeks
Population: as for outcome 20
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) | Atorvastatin 10, 20, 40, or 80 mg (Pooled)
Number analyzed (Participants) | 732 | 1607
Percentage of Participants | 59.6 | 45.9
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) vs Atorvastatin 10, 20, 40, or 80 mg (Pooled); Test type: Superiority or Other; Miettinen and Nurminen; Difference in Percentage = 13.7, 95% CI 2-sided [9.4 to 18.0]

22. Secondary Outcome: Percentage of Participants Who Experience at Least 1 Laboratory Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. A laboratory AE was an AE reported as a result of a laboratory assessment or test.
Time Frame: up to 14 weeks
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) | Atorvastatin 10, 20, 40, or 80 mg (Pooled)
Number analyzed (Participants) | 732 | 1607
Percentage of Participants | 5.2 | 5.9
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) vs Atorvastatin 10, 20, 40, or 80 mg (Pooled); Test type: Superiority or Other; Miettinen and Nurminen; Difference in Percentage = -0.7, 95% CI 2-sided [-2.6 to 1.4]

23. Secondary Outcome: Percentage of Participants Who Were Discontinued From the Study Due to a Clinical AE
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. A clinical AE was an AE reported as a result of a clinical examination or reported by the participant. Participants who were discontinued from the study due to a clinical AE were recorded.
Time Frame: up to 14 weeks
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) | Atorvastatin 10, 20, 40, or 80 mg (Pooled)
Number analyzed (Participants) | 732 | 1607
Percentage of Participants | 16.5 | 4.9
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) vs Atorvastatin 10, 20, 40, or 80 mg (Pooled); Test type: Superiority or Other; Miettinen and Nurminen; Difference in Percentage = 11.7, 95% CI 2-sided [8.9 to 14.7]

24. Secondary Outcome: Percentage of Participants Who Were Discontinued From the Study Due to a Laboratory AE
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. A laboratory AE was an AE reported as a result of a laboratory assessment or test. Participants who were discontinued from the study due to a laboratory AE were recorded.
Time Frame: up to 14 weeks
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) | Atorvastatin 10, 20, 40, or 80 mg (Pooled)
Number analyzed (Participants) | 732 | 1607
Percentage of Participants | 0.7 | 0.7
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) vs Atorvastatin 10, 20, 40, or 80 mg (Pooled); Test type: Superiority or Other; Miettinen and Nurminen; Difference in Percentage = -0.1, 95% CI 2-sided [-0.8 to 0.9]

25. Secondary Outcome: Percentage of Participants Who Experience at Least 1 Hepatitis-related Clinical AE
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. Hepatitis-related AEs were identified by a collective review using the following pre-specified set of preferred terms: cholestasis, hepatic necrosis, hepatocellular damage, cytolytic hepatitis, hepatitis, hepatomegaly, jaundice, hepatic failure, hepatitis cholestatic, jaundice cholestatic, hepatitis fulminant, hyperbilirubinaemia, jaundice hepatocellular, ocular icterus, yellow skin, hepatic function abnormal, acute hepatic failure, subacute hepatic failure, hepatitis acute, hepatitis toxic, hepatotoxicity, and mixed hepatocellular-cholestatic injury.
Time Frame: up to 14 weeks
Population: as for outcome 20
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) | Atorvastatin 10, 20, 40, or 80 mg (Pooled)
Number analyzed (Participants) | 732 | 1607
Percentage of Participants | 0.0 | 0.1
Statistical Analysis 1: Comparison: MK-0524B 2g/20 mg or MK-0524B 2g/40mg (Pooled) vs Atorvastatin 10, 20, 40, or 80 mg (Pooled); Test type: Superiority or Other; p = 0.4997, Miettinen and Nurminen; Difference in Percentage = -0.1, 95% CI 2-sided [-0.4 to 0.5]

ADVERSE EVENTS:
Time Frame: up to 14 weeks
Groups:
- MK-0524B 2g/40 mg: Co-administration of one tablet of MK-0524A 1g + one tablet of simvastatin 20 mg for 4 weeks, then co-administration of two tablets of MK-0524A 1g + simvastatin 40 mg for 8 weeks
Arm/Group | MK-0524B 2g/20 mg | MK-0524B 2g/40 mg | Atorvastatin 10 mg | Atorvastatin 20 mg | Atorvastatin 40 mg | Atorvastatin 80 mg
Serious Adverse Events (participants affected / at risk) | 3/297 | 8/435 | 3/298 | 5/439 | 3/437 | 7/433
Other Adverse Events (participants affected / at risk) | 71/297 | 136/435 | 25/298 | 27/439 | 31/437 | 35/433
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0524B 2g/20 mg (N=297) | MK-0524B 2g/40 mg (N=435) | Atorvastatin 10 mg (N=298) | Atorvastatin 20 mg (N=439) | Atorvastatin 40 mg (N=437) | Atorvastatin 80 mg (N=433)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angle closure glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Device malfunction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0524B 2g/20 mg (N=297) | MK-0524B 2g/40 mg (N=435) | Atorvastatin 10 mg (N=298) | Atorvastatin 20 mg (N=439) | Atorvastatin 40 mg (N=437) | Atorvastatin 80 mg (N=433)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 13 (14) | 15 (16) | 15 (15) | 18 (19) | 15 (18)
Pruritus (Skin and subcutaneous tissue disorders) | 16 (23) | 28 (33) | 3 (3) | 3 (4) | 2 (2) | 1 (1)
Flushing (Vascular disorders) | 57 (67) | 102 (120) | 7 (7) | 11 (13) | 12 (12) | 19 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.